CLINICAL TRIAL: NCT05278702
Title: Autonomic Nervous System Dysfunction in Patients With End-stage Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Faitatzidou Danai, PhD candidate, Aristotle University Of Thessaloniki
Other Study IDs: ΔΔ4844
Record Dates: First submitted 2022-02-23; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Kidney Failure, Chronic
Keywords: hemodialysis; autonomic nervous system; peritoneal dialysis; end-stage kidney disease; heart rate variability
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hemodialysis
- peritoneal dialysis

SUMMARY:
The prevalence of autonomic nervous system (ANS) dysfunction in patients with end-stage kidney disease (ESKD) is considered to be increased. The uraemic environment, as well as the high incidence of comorbid conditions affecting the ANS function (e.g. diabetes mellitus, autoimmune and degenerative neurological diseases), have been proposed to cause important alterations in ANS function. The vast majority of evidence on the prevalence of ANS dysfunction in ESKD patients is derived from small studies elaborating simple methodology. Noteworthy, with the exception of a study in 27 hemodialysis patients which assessed ANS function before and after dialysis in relation to left ventricular filling pressures, and a 2005 Dutch study in 21 patients whether or not they had hypotension during dialysis, no other study used advanced methods to analyze heart rate or blood pressure variability from beat-to-beat recordings, such as this study. In addition, there is no study so far investigating possible changes in the ANS function per dialysis session. Finally, to the best of our knowledge, this is the first work evaluating possible differences in ANS function in hemodialysis compared with peritoneal dialysis individuals.

DETAILED DESCRIPTION:
This is an observational study performed in the Department of Nephrology, Hippokration Hospital, Thessaloniki, Greece. For the purposes of this study, adult patients (>18 years) with ESKD being treated with hemodialysis (HD) (on standard thrice-weekly HD treatment) or peritoneal dialysis (PD) for at least 3 months, fulfilling the inclusion/exclusion criteria were invited to participate. PD and HD patients will be matched by a blinded member of our team based on age, gender and dialysis vintage (i.e. the duration of time after the point they started renal replacement therapy for ESRD) in a 1:1 ratio. All included patients signed a written informed consent form. The study protocol was approved by the Ethics Committee of the School of Medicine, Aristotle University of Thessaloniki. All procedures and evaluations are performed according to the Declaration of Helsinki 2013 Amendment.

Evaluation of participants includes the recording of demographics and anthropometric characteristics, medical history, concomitant medications and dialysis-related parameters, as well as physical examination and venous blood sampling for routine laboratory tests. Participants are instructed to visit the Department one hour before the programmed follow-up visit at their unit (PD patients); HD patients are instructed to visit the Department on 2 consecutive days (mid-week dialysis day and the corresponding dialysis-off day). All procedures are performed in a room with an ambient temperature of 23-24oC. Firstly, participants are oriented and familiarized with the experimental procedures and are prepared for the hemodynamic and cardiovascular examinations. Continuous beat-by-beat BP and heart rate are monitored using finger photoplethysmography (Finometer PRO, Finapres Medical Systems, Amsterdam, the Netherlands) throughout the protocol. An inflatable cuff is placed on the middle finger of the non-access hand maintained at heart level. After a 5-min rest, all participants underwent a mental task (countdown from 100 to 0 by 7, performed twice), an orthostatic test (5 min with the patient at the supine position followed by 5 min with the patient in upright position), and a mild physical task [3-minute submaximal handgrip exercise test (set of 30 s exercise at 35% MVC with 3 s rest] (K-Force, K-invent). At the completion of the exercise protocol, the Rate of Perceived Exertion (RPE) is assessed using the Borg scale.

For data analysis, beat-by-beat SBP and DBP will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands). From pulse pressure profiles, beat-by-beat heart rate (HR) and stroke volume (SV, ml) will be computed, using the Modelflow method; cardiac output (L/min) and systemic vascular resistance (SVR, mmHg.s/mL), will also be computed using Beatscope. HRV analysis will be performed with the HRV Analysis software Kubios (version 3.3.1, Kubios Oy, 2019) by the same researcher to eliminate inter-observer variability. R-R interval series will be checked for ectopic beats or artifacts. The root mean square of successive differences (RMSSD) between the coupling intervals of adjacent R-R intervals will be used as a parasympathetic activity index. Baroreceptor sensitivity (ms/mmHg) will be assessed by examining the spontaneous fluctuations in the blood pressure as assessed by the cross-correlation method using the Beatscope 1a software).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* ESKD individuals treated with either hemodialysis (standard thrice weekly schedule) or peritoneal dialysis for at least 3 months
* Provision of informed written consent

Exclusion Criteria:

* Antihypertensive treatment modifcation during one month prior to study enrollment
* Modification of treatment for neurological disorders one month prior to study enrollment
* Active malignant disease or other comorbidity with poor prognosis
* History of neurological disorders (e.g. Parkinson's disease, multiple sclerosis, etc) that cause primary ANS dysfunction
* History of ANS dysfunction secondary to diabetes mellitus, amyloidosis, autoimmune disorders, etc.
* Active infection or relevant inter-current illness.
* History of drug or alcohol abuse or severe mental disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESKD individuals treated with either hemodialysis (standard thrice weekly schedule) or peritoneal dialysis
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference in the root mean square of successive R-R differences [RMSSD (ms)] parameter of heart rate variability during the mental arithmetic test between the examination during the dialysis session and the examination in the out-of-dialysis day | Baseline
  The root mean square of successive differences (RMSSD) between the coupling intervals of adjacent R-R intervals will be used as a parasympathetic activity index. RMSSD will be calculated with the HRV Analysis software Kubios (version 3.3.1, Kubios Oy, 2019)

SECONDARY OUTCOMES:
The difference in baroreceptor-sensitivity (ms/mmHg) during mental-arithmetic-test between examination during the session and examination in the out-of-dialysis day. | Baseline
  Baroreceptor sensitivity (ms/mmHg) will be assessed by examining the spontaneous fluctuations in the blood pressure as assessed by the cross-correlation method using the Beatscope 1a software).
The difference in stroke-volume (ml) during mental-arithmetic-test between examination during the session and examination in the out-of-dialysis day. | Baseline
  Beat-by-beat stroke volume (ml) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in cardiac-output (L/min) during mental-arithmetic-test between examination during the session and examination in the out-of-dialysis day | Baseline
  Beat-by-beat cardiac output (L/min) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands).
The difference in total-peripheral-resistance during mental-arithmetic-test between examination during the session and examination in the out-of-dialysis day. | Baseline
  Beat-by-beat total peripheral resistance (mmHg.s/mL) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in both SBP and DBP (mmHg) during mental-arithmetic-test between examination during the session and examination in the out-of-dialysis day. | Baseline
  Beat-by-beat SBP and DBP will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in in the root mean square of successive R-R differences [RMSSD (ms)] parameter of heart rate variability during the handgrip test between dialysis session start and session end. | Baseline
  The root mean square of successive differences (RMSSD) between the coupling intervals of adjacent R-R intervals will be used as a parasympathetic activity index. RMSSD will be calculated with the HRV Analysis software Kubios (version 3.3.1, Kubios Oy, 2019)
The difference in baroreceptor sensitivity (ms/mmHg) during the handgrip test between dialysis session start and session end. | Baseline
  Baroreceptor sensitivity (ms/mmHg) will be assessed by examining the spontaneous fluctuations in the blood pressure as assessed by the cross-correlation method using the Beatscope 1a software).
The difference in cardiac output (L/min) during the handgrip test between dialysis session start and session end. | Baseline
  Beat-by-beat cardiac output (L/min) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in total peripheral resistance during the handgrip test between dialysis session start and session end. | Baseline
  Beat-by-beat total peripheral resistance (mmHg.s/mL) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in both SBP and DBP (mmHg) during the handgrip test between dialysis session start and session end. | Baseline
  Beat-by-beat SBP and DBP will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in stroke volume (ml) during the handgrip test between dialysis session start and session end. | Baseline
  Beat-by-beat stroke volume (ml) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in in the root mean square of successive R-R differences [RMSSD (ms)] parameter of heart rate variability during the orthostatic test between dialysis session start and session end | Baseline
  The root mean square of successive differences (RMSSD) between the coupling intervals of adjacent R-R intervals will be used as a parasympathetic activity index. RMSSD will be calculated with the HRV Analysis software Kubios (version 3.3.1, Kubios Oy, 2019)
The difference in baroreceptor sensitivity (ms/mmHg) during the orthostatic test between dialysis session start and session end. | Baseline
  Baroreceptor sensitivity (ms/mmHg) will be assessed by examining the spontaneous fluctuations in the blood pressure as assessed by the cross-correlation method using the Beatscope 1a software).
The difference in stroke volume (ml) during the orthostatic test between dialysis session start and session end. | Baseline
  Beat-by-beat stroke volume (ml) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in cardiac output (L/min) during the orthostatic test between dialysis session start and session end. | Baseline
  Beat-by-beat cardiac output (L/min) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in the total peripheral resistance during the orthostatic test between dialysis session start and session end. | Baseline
  Beat-by-beat total peripheral resistance (mmHg.s/mL) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in both SBP and DBP (mmHg) during the orthostatic test between dialysis session start and session end. | Baseline
  Beat-by-beat SBP and DBP will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in in the root mean square of successive R-R differences [RMSSD (ms)] parameter of heart rate variability during the handgrip test between hemodialysis and peritoneal dialysis patients:. | Baseline
  The root mean square of successive differences (RMSSD) between the coupling intervals of adjacent R-R intervals will be used as a parasympathetic activity index. RMSSD will be calculated with the HRV Analysis software Kubios (version 3.3.1, Kubios Oy, 2019)
The difference in the baroreceptor sensitivity (ms/mmHg) during the handgrip test between hemodialysis and peritoneal dialysis patients:. | Baseline
  Baroreceptor sensitivity (ms/mmHg) will be assessed by examining the spontaneous fluctuations in the blood pressure as assessed by the cross-correlation method using the Beatscope 1a software).
The difference in the stroke volume (ml) during the handgrip test between hemodialysis and peritoneal dialysis patients:. | Baseline
  Beat-by-beat stroke volume (ml) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in the total peripheral resistance during the handgrip test between hemodialysis and peritoneal dialysis patients:. | Baseline
  Beat-by-beat total peripheral resistance (mmHg.s/mL) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in the cardiac output (L/min) during the handgrip test between hemodialysis and peritoneal dialysis patients. | Baseline
  Beat-by-beat cardiac output (L/min) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in both SBP and DBP (mmHg) during the handgrip test between hemodialysis and peritoneal dialysis patients. | Baseline
  Beat-by-beat SBP and DBP will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in in the root mean square of successive R-R differences [RMSSD (ms)] parameter of heart rate variability during the orthostatic test between hemodialysis and peritoneal dialysis patients. | Baseline
  The root mean square of successive differences (RMSSD) between the coupling intervals of adjacent R-R intervals will be used as a parasympathetic activity index. RMSSD will be calculated with the HRV Analysis software Kubios (version 3.3.1, Kubios Oy, 2019)
The difference in baroreceptor sensitivity (ms/mmHg) during the orthostatic test between hemodialysis and peritoneal dialysis patients. | Baseline
  Baroreceptor sensitivity (ms/mmHg) will be assessed by examining the spontaneous fluctuations in the blood pressure as assessed by the cross-correlation method using the Beatscope 1a software).
The difference in cardiac output (L/min) during the orthostatic test between hemodialysis and peritoneal dialysis patients. | Baseline
  Beat-by-beat cardiac output (L/min) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in total peripheral resistance during the orthostatic test between hemodialysis and peritoneal dialysis patients. | Baseline
  Beat-by-beat total peripheral resistance (mmHg.s/mL) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in stroke volume (ml) during the orthostatic test between hemodialysis and peritoneal dialysis patients. | Baseline
  Beat-by-beat stroke volume (ml) will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)
The difference in both SBP and DBP (mmHg) during the orthostatic test between hemodialysis and peritoneal dialysis patients. | Baseline
  Beat-by-beat SBP and DBP will be averaged per testing session and exported using the Beatscope software (version 1.a, Finapres Medical Systems, Amsterdam, the Netherlands)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Hippokration Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Savica V, Musolino R, Di Leo R, Santoro D, Vita G, Bellinghieri G. Autonomic dysfunction in uremia. Am J Kidney Dis. 2001 Oct;38(4 Suppl 1):S118-21. doi: 10.1053/ajkd.2001.27418. PMID 11576936
- [Background] Kamal A. Effect of hemodialysis on autonomic dysfunction in patients with chronic renal failure - biomed 2009. Biomed Sci Instrum. 2009;45:280-5. PMID 19369776
- [Background] Galiatsatos P, Parakh K, Monti J, Thavarajah S, Aneke-Ogbu H, Watson A, Kim D, Wang NY, Shafi T, Silber HA. A finger photoplethysmography waveform during the valsalva maneuver detects changes in left heart filling pressure after hemodialysis. BMC Nephrol. 2015 Aug 14;16:138. doi: 10.1186/s12882-015-0135-0. PMID 26272208
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Parati G, Casadei R, Groppelli A, Di Rienzo M, Mancia G. Comparison of finger and intra-arterial blood pressure monitoring at rest and during laboratory testing. Hypertension. 1989 Jun;13(6 Pt 1):647-55. doi: 10.1161/01.hyp.13.6.647. PMID 2500393
- [Background] Dipla K, Kousoula D, Zafeiridis A, Karatrantou K, Nikolaidis MG, Kyparos A, Gerodimos V, Vrabas IS. Exaggerated haemodynamic and neural responses to involuntary contractions induced by whole-body vibration in normotensive obese versus lean women. Exp Physiol. 2016 Jun 1;101(6):717-30. doi: 10.1113/EP085556. PMID 27061448
- [Background] Westerhof BE, Gisolf J, Stok WJ, Wesseling KH, Karemaker JM. Time-domain cross-correlation baroreflex sensitivity: performance on the EUROBAVAR data set. J Hypertens. 2004 Jul;22(7):1371-80. doi: 10.1097/01.hjh.0000125439.28861.ed. PMID 15201554
- [Derived] Faitatzidou D, Dipla K, Theodorakopoulou MP, Koutlas A, Tsitouridis A, Dimitriadis C, Pateinakis P, Zafeiridis A, Papagianni A, Jadoul M, Sarafidis P. Heart rate variability at rest and in response to stress: Comparative study between hemodialysis and peritoneal dialysis patients. Exp Biol Med (Maywood). 2023 Oct;248(20):1745-1753. doi: 10.1177/15353702231198081. Epub 2023 Nov 2. PMID 37916412